CLINICAL TRIAL: NCT06532097
Title: Initial Effect Size Estimation of a Smartwatch-based Intervention for Physical and Behavioral Activation in Depressed Patients: a Pilot-study
Brief Title: Initial Effect Size Estimation of a Smartwatch-based Intervention for Physical and Behavioral Activation in Depressed Patients
Status: Completed | Type: Observational
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Sponsor
Other Study IDs: MaxPlanckIP
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention group: Group of patients that received the digital intervention
  Interventions: Behavioral: Physical and behavioral smartwatch-based activation
- Retrospective control group: Retrospectively collected group of patients from earlier versions (amendments) of the study who filled out the PHQ-9 twice with a certain interval (and were offered the intervention at a later time-point)

INTERVENTIONS:
Behavioral: Physical and behavioral smartwatch-based activation — We used smartwatches to provide an interactive tool for delivering a mixed intervention of physical and behavioral activation, with the former addressing physical activity level and the latter pleasant activities including and beyond physical activity (e.g., social, relaxing activities). Moreover, given the relationship with physical activity level, we additionally incorporated digital insomnia exercises that have also shown large effects in the amelioration of depression.
  Groups: Intervention group

SUMMARY:
It is well known that physical activity interventions have a robust, if small-to-moderate effect on the amelioration of chronic diseases, including major depressive disorder (MDD) (Singh et al. 2023). At the same time, behavioral activation is one of the most effective components of digital cognitive-behavioral therapy for depression (Furakawa et al. 2021). Here we leveraged smartwatches to provide an interactive tool for delivering a mixed intervention of physical and behavioral activation, with the former addressing physical activity level and the latter pleasant activities including and beyond physical activity (e.g., social, relaxing activities). Moreover, given the relationship with physical activity level, we additionally incorporated digital insomnia exercises that have also shown promising effects in the amelioration of depression. Our primary aim was to estimate the effects of our digital smartwatch-based intervention in a small sample of depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* Written consent for voluntary study participation
* Between 18 and 65 years of age
* Current diagnosis of a single episode of mild to moderate depressive disorder without psychotic symptoms, according to ICD-10 (F32.0, F32.1)
* Internet access and email address to answer electronic questionnaires
* Ability to read German

Exclusion Criteria:

* Acute suicidality
* Pregnancy and breastfeeding
* Currently undergoing psychological treatment
* Current use of psychotropic medication
* Neurological or internal medical disease
* Diagnosis of a severe major depression or dysthymia according to ICD-10 (F32.2, F32.3, F33.2, F33.3, F34.1)
* Diagnosis of a psychotic disorder according to ICD-10 (F20-F29) in the life history
* Diagnosis of a bipolar disorder according to ICD-10 (F31) in life history
* Acute substance abuse (e.g., drug use or excessive alcohol and nicotine use)
* Diagnosis of dissociative disorder (F44) in life history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unmedicated, depressed patients (mildly or moderately depressed).
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
PHQ-9 | pre to post: 12 weeks
  Patient Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Victor Spoormaker, PhD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Depending on privacy regulation (removal of all connections to personal identifiers), the aim is to make the primary readout scores available.